CLINICAL TRIAL: NCT01606033
Title: Psychological and Emotional Impacts of Participation in Oncologic Clinical Trials
Brief Title: Study of Stress and Life Quality of Patients Participating in Clinical Trials Versus Patients Non Participating
Acronym: IPSY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IPSY 0905
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Metastatic Neoplasm; Recurrent Hematologic Cancer
Keywords: stress; Life quality; adjustment strategy; receiving an antitumor treatment; within a clinical trial (case); according to a standard treatment (control)
MeSH Terms: conditions — Neoplasm Metastasis; Hematologic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- phase II non randomized study (Other): phase II non randomized study, "Case" : 40 patients description of patients feeling by questionnaires :
  * Anxiety and depression questionnaire, life quality questionnaire, adjustment strategy questionnaire, emotional regulation questionnaire, satisfaction Survey
  * understanding of the implications of participating in a clinical trial
  Interventions: Other: questionnaires; Other: questionnaire
- blind randomized phase II or III study (Other): blind randomized phase II or III study: "control" : 40 patients description of patients feeling by questionnaires :
  * Anxiety and depression questionnaire, life quality questionnaire, adjustment strategy questionnaire, emotional regulation questionnaire, satisfaction Survey
  * understanding of the implications of participating in a clinical trial
  Interventions: Other: questionnaires; Other: questionnaire
- open randomized phase II or III study (Other): open randomized phase II or III study : 40 patients description of patients feeling by questionnaires : Anxiety and depression questionnaire, life quality questionnaire, adjustment strategy questionnaire, emotional regulation questionnaire, satisfaction Survey
  -understanding of the implications of participating in a clinical trial
  Interventions: Other: questionnaires; Other: questionnaire
- receiving standard treatment (Other): receiving standard treatment : 120 patients description of patients feeling by questionnaires :
  -understanding of the implications of participating in a clinical trial
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — Anxiety and depression questionnaire, life quality questionnaire, adjustment strategy questionnaire, emotional regulation questionnaire, satisfaction survey
Other: questionnaire — understanding of the implications of participating in a clinical trial
  Arms: blind randomized phase II or III study; open randomized phase II or III study; phase II non randomized study

SUMMARY:
This study aims to assess anxiety/depression and life quality of patients included in clinical trials versus patients treated in a standard way.

DETAILED DESCRIPTION:
This study aims to assess anxiety/depression and life quality of patients included in clinical trials versus patients treated in a standard way A case-control study

ELIGIBILITY:
Inclusion Criteria:

* patient with solid tumor or recurrent hematologic cancer, treated by chemotherapy or targeted therapy evaluated every 2 or 3 cycles; except for clinical trials associating non drug treatment (radiotherapy, surgery...)
* subject to a 1st, 2nd or 3rd line of antitumor treatment

  * a phase 2 open labeled study,
  * a phase 2 or 3 blind randomised study,
  * a phase 2 or 3 open randomised study,
  * a standard treatment non participating to a clinical trial
* male or female patients ≥ 18 years of age
* karnovsky ≥ 70 % or OMS ≤ 2
* recovered from prior toxicities
* social security covered
* written informed consent given

Exclusion Criteria:

* psychiatric disorders, receiving psychotropic treatment
* physical or psychological issues
* forbidden to be included in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-03; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
assess and compare stress and life quality of patients participating to a clinical trial vs patients treated a standard way | 4 years
  quality of life questionnaire (QLQ C30) Anxiety and depression questionnaire (HADS)

SECONDARY OUTCOMES:
evaluate links between using adjustment therapy and emotional regulation, and emotional and psychological experience of patients facing one or another situation | 4 years
  adjustment therapy questionnaire (WCC) emotional regulation questionnaire (DERS 24)
measure and compare variation in time of psychological and emotional consequences during treatment | 5 years
  emotional regulation (DERS 24)
measure the level of knowledge on the implications of participating in a clinical trial (case) | 5 years
  assess impact of it on psychological and emotional experience

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie CLISANT, Study Director — Oscar Lambret Center
Locations (8):
- France (8):
  - Oscar Lambret Center, Lille, Hauts-de-France
  - Paul PAPIN Center, Angers
  - François Baclesse Center, Caen
  - CHOLET Hospital, Cholet
  - Georges-François LECLERC Center, Dijon
  - Léon BERARD Center, Lyon
  - Val D'AURELLE Center, Montpellier
  - Jean GODINOT Institut, Reims

IPD SHARING:
Plan to Share IPD: No